CLINICAL TRIAL: NCT04752592
Title: Evaluation of the Feasibility, Accuracy, and Effect of a Rapid Point-of-Care Serological Triage Test for Active TB (SeroSelectTB) in High Burden, HIV-endemic African Settings: a Multi-centre, Parallel-group, Randomised, Controlled Trial
Brief Title: Evaluation of a Rapid Point-of-Care Serological Triage Test for Active TB
Acronym: SeroSelectTB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Institute of Public Health (Other Government)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); University of Stellenbosch (Other); Kilimanjaro Christian Medical University College (Unknown); Armauer Hansen Research Institute, Ethiopia (Other); Lateral Flow Laboratories (Pty) Ltd (Unknown); InVivo BioTech Services GmbH (Unknown); Aether Dynamics Consulting & Trading GmbH (Unknown); E-MEDDIA (Unknown); KNCV Tuberculosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 19/10773
Record Dates: First submitted 2021-02-04; First posted 2021-02-12 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Tuberculosis, Pulmonary
Keywords: Tuberculosis; Rapid diagnostics; Triage test; Diagnostic delay; Low-income countries; Africa
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SeroSelectTB (Experimental): The participants in this arm, after providing informed concent, will be tested using the SeroSelectTB rapid assay.
  Interventions: Diagnostic Test: SeroSelectTB rapid TB test
- Standard of Care (No Intervention): The participants in this arm, after providing informed consent, will receive the established standard of care.

INTERVENTIONS:
Diagnostic Test: SeroSelectTB rapid TB test — The SeroSelectTB test is a rapid blood-based immunochemical lateral flow assay for the detection of active tuberculosis.
  Arms: SeroSelectTB

SUMMARY:
The performance of a new triage test for active tuberculosis (TB), SeroSelectTB, will be qualified in multi-centre randomised controlled trials at health-posts in South Africa, Tanzania and Ethiopia. Cost effectiveness evaluations will be conducted to support a value proposition to stakeholders and regulatory authorities, and to support commercialization requirements.

Consenting adults will provide blood and saliva samples for screening by SeroSelectTB, and sputum collected for routine TB diagnosis by the health services. Clinical and sociodemographic information will be collected.

A reliable rapid test will make it possible to identify and selectively treat those with active TB at the local healthcare level. The expected impact includes accurate same-day diagnosis of patients with active TB, reduction of diagnostic delay and TB transmission, and diagnostic cost-savings for patients and healthcare systems in high TB-burden countries.

DETAILED DESCRIPTION:
Purpose: Worldwide over 15 million persons live with active TB. While the prevalence of latent TB is very high, only disease, and not latent infection, is treated in most high burdened countries.

A rapid triage test for detection of active TB, which can identify symptomatic individuals who require confirmatory diagnostic investigation, is a global priority for TB control. A rapid triage test can drastically reduce the burden on health systems and patients, and reduce diagnostic delay by expediting referral, confirmatory testing and timely commencement of adequate treatment. Triage tests, which may utilise point- of-care rapid lateral flow (LF) platforms, offer a promising alternative to conventional methods for TB diagnosis (i.e. smear microscopy and culture). However, the lack of accurate TB biomarkers has stalled the development of serological assays that meet the World Health Organization (WHO)-defined criteria for a triage test.

As an alternative, a rapid molecular diagnostic tool, maned Xpert and Xpert Ultra MTB/RIF, which accurately detects active TB, has been introduced in many countries as a replacement for smear microscopy and culture. However, Xpert/Ultra is not suited for use at health-posts without electricity or laboratory facilities, where the majority of patients present. In addition, the affordability of scaling-up Xpert is of concern in high TB-burden countries, where it could consume 20-80% of national TB budgets.

Therefore, to control the emergence and spread of antibiotic resistant TB in a cost-effective manner, there is an urgent need for a rapid, inexpensive triage test that can detect active TB at health-posts level and expedite referral to facilities supporting molecular diagnostics. An ideal cost-effective triage test should be as sensitive as Xpert and cost less than US $5 to reduce total diagnostic costs by 30-40%, potentially saving national TB programmes US $36 million/year.

The expected outcome of this project, the implementation of a triage test that will detect active TB at a low diagnostic cost, and expedite persons with TB-indicative symptoms to centralized healthcare facilities, will be beneficial irrespective of age and gender of patients. In addition, SeroSelectTB is sensitive among adults co- infected with TB/HIV.

Primary objective of field trial is to evaluate the diagnostic delay, measured as the time from TB diagnostic to TB treatment initiation between two groups of patients: those who were screened with SeroSelectTB triage test compared to patients who received the standard of care.

Persons with reactive SeroSelectTB test results will be referred for same-day confirmatory Xpert testing and treatment.

Secondary objectives are:

* To describe SeroSelectTB performance in field conditions, including sensitivity and specificity, positive and negative predictive values in the study populations.
* Collect blood and saliva samples from all consenting participants and create national biobanks, which will facilitate biological samples exchange and sharing with third parties for future research.
* Assess the added-value of using SeroSelectTB in healthcare systems in South Africa, Tanzania and Ethiopia through cost-effectiveness evaluation and inform international and national TB prevention programmes stakeholders.

Study design: This is an interventional, a multi-centre, two parallel-group, randomised, controlled field trial conducted in three countries: The South African Republic, United Republic of Tanzania, and Republic of Ethiopia.

In the interventional arm participants will be screened using SeroSelectTB rapid triage test, and in the case of positive SeroSelectTB test results, will be referred to TB confirmation diagnostics at the referral centre where TB diagnosis will be confirmed by Xpert/Ultra molecular diagnostics. In the standard of care arm patients will receive usual TB diagnostics: microbiology (culture-confirmed diagnostics) and/or microscopy (sputum smear-based diagnostics).

At inclusion, participants will be blinded to which diagnostic arm they are randomized: SeroSelectTB or standard of care arm. Healthcare workers performing the diagnostic test will not be blinded since it is unattainable to conceal if they are performing a microscopy/culture-based diagnostics or hand-held SeroSelectTB test. Lab technicians at Lateral Flow Laboratories, South Africa, and the National Institute of Health and the Environment (RIVM), the Netherlands will be blinded to patients' allocation when performing quality control analyses.

Recruitment strategy and retention: An information leaflet and booklet addressing 'Myths and Facts' about TB diagnostic testing and the clinical trial, respectively, have been produced and translated from English to Kiswahili, Amharic, isiXhosa and Afrikaans. This information will be submitted to ethics committees for approval, and be used for public dissemination as a community engagement tool and given to every study participant.

Healthcare facilities and clinical centres involved in this study have access to more than 7,000 suspected TB cases per year, which ensures a large enough population to identify patients with active pulmonary TB disease.

Loss to follow-up will be minimized by involving the community upfront through our planned community engagement plan, performing follow-up interviews with patients on TB treatment (DOTs - directly observed therapy - patients will be followed-up by data collection regarding their treatment), and/or conducting home visits.

Recruitment site selection: Healthcare facilities and centres were selected based on reported high TB burden and previous experience with clinical and field TB trials. Annually, more than the double of confirmed TB cases are reported in the selected sites, which makes recruitment of needed number of cases (N=123) over two years' time feasible.

Study safety: This trial does not contain any experimental intervention that will influence patients care. Collection of biological samples will be in accordance with WHO guidelines on blood sampling for research purposes.

Study monitoring and data management: A written contractual agreement ('Consortium Agreement') will be signed by the consortium partners, and specific Clinical Trial Agreements will be signed by the Norwegian Institute of Public Health (NIPH) and clinical trial centers: Stellenbosch University, South African Republic, Kilimanjaro Christian Medical University College, United Republic of Tanzania, and Armauer Hansen Research Institute, Republic of Ethiopia, before the study start. A primary investigator (PI) at the trial center will be responsible for reaching milestones, informing work package (WP) and consortium Steering Committee (SC) leaders on progress, and keeping accounts as defined in project guidelines.

On-site and in-house monitoring of trial data and protocol compliance will be performed according to study analysis protocol, written study plans and standard operating procedures (SOPs). An independent Data Monitoring Committee (DMC) composed of study site principal investigators (PIs), individuals with relevant expertise (e.g. data management and/or clinical background), and a statistician from NIPH will report directly to the SC. The role of DMC is to monitor data collection, data integrity and project timelines related to data collection. In addition, Field Evaluation Trial Committee (FETC), formed by local healthcare workers and clinicians, will be responsible for trial sites patients' safety and integrity. The FETC will closely work with DMC, and report to the SC.

A risk-based approach to monitoring will be used. A secured cloud system will be used to register screened participants, randomization and assign to a trial arm. Data management, including cloud system design and maintenance, data cleaning, creation of listings for in-house monitoring, developing randomisation schedule, progress reports, Statistical Analysis Plan development, tables, figures, and presentations, and evaluation of primary and secondary end points, will be overseen by DMC and FETC.

The study sponsor will host the database and maintain the oversight over recruitment, protocol compliance, study conduct, data correctness and integrity. Monitoring (on-site and remotely) and data management will be in the remit of DMC and FETC.

No data whatsoever will be generated in the European Union (EU) or Norway, or stored on a server in the EU or Norway. Data will be stored solely on the institutional servers at our partner institutions in South Africa, Tanzania, and Ethiopia as required by institutional and national guidelines. To ensure data protection we guarantee that:

* Data extracted from the SeroSelectTB case report form entered into and stored on national servers in South Africa, Ethiopia, and Tanzania will be anonymized.
* A one-way random algorithm will automatically scramble data rows before data is shared with the project researchers.
* Data cannot be traced back to the source/participant.
* Personal identifier information is protected and available only to the national health services in South Africa, Ethiopia, and Tanzania as required by national guidelines.
* Data made available for analysis (shared with project researchers) will be provided f.ex. on Excel spread sheets without the unique participant codes.
* The Excel data files will be destroyed after analysis and publication of results.

Sub-Studies:

SeroSelectTB will also biobank blood specimens to evaluate the diagnostic accuracy of concise blood transcriptional signatures in symptomatic patients, such as in one of its ancillary studies, RADIANT (https://www.sun.ac.za/english/faculty/healthsciences/Molecular_Biology_Human_Genetics/clinical_mycobacteriology_epidemiology/Pages/RADIANT.aspx).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Informed Consent Form signed
* Unwell, suspected to have TB or pneumonia

Exclusion Criteria:

* Currently receiving TB treatment
* On TB treatment past 30 days or more, or last dose less than 1 month before enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9097 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
To determine the impact of SeroSelectTB on health systems' diagnostic delay in Ethiopia, Tanzania and South Africa. | The time points will be measure from the data of SeroSelectTB test or standard-of-care until the start of treatment (when active TB is diagnosed). Participants receiving TB therapy will be followed for 6 months according to national routines.
  Our hypothesis is that the use of a rapid triage assay at patients' first encounter with the healthcare system will, when compared to the standard-of-care, reduce time to TB diagnosis.
  The assessment of the primary objective will be based on two complementary measures: primary measure is time to diagnosis (measured in days), and secondary measure is time to treatment (measured in days).

SECONDARY OUTCOMES:
To describe SeroSelectTB performance in field conditions, including sensitivity and specificity, and positive and negative predictive values, in the study populations. | Investigations will be performed during the intervention.
  Test accuracy will be documented through bench-based evaluations at partner institutions in Cape Town and through external quality control investigations at RIVM.
Evaluate cost-effectiveness of SeroSelectTB. | Cost effectiveness will be determined at year 6.
  The overall cost of TB diagnosis, treatment and care by 1) implementing a new rapid triage test at peripheral healthcare facilities and 2) standard-of-care at peripheral healthcare facilities will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Grant Theron, PhD, Principal Investigator — University of Stellenbosch; Balthazar Nyombi, PhD, Principal Investigator — Kilimanjaro Christian Medical Center University; Kidist Bobosha, PhD, Principal Investigator — Armauer Hansen Research Institute; Carol Holm-Hansen, PhD, Principal Investigator — Norwegian Institute of Public Health
Locations (3):
- Amhara region, Bahir Dar, Ethiopia
- Stellenbosch University Clinics, Cape Town, Western Cape, South Africa
- Kilimanjaro region, Tanzania, Moshi, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
Only the documents below will be shared. No data with personal identifiers will be shared, all shared data that will be analysed will be anonymized and scrambled.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The anonymized data will be available for two years after the date of final publication.
Access Criteria: Interested parties should directly contact the principle investigators to request access and adhere to the institutional and national regulations for data sharing.
URL: http://www.fhi.no

REFERENCES:
- See also: Project website — http://www.seroselecttb.org
- Available data/document: Study Protocol — https://www.seroselecttb.org/resources